CLINICAL TRIAL: NCT03397030
Title: Impact of a Home-based Exercise Program on Prognostic Biomarkers in Men With Prostate Cancer
Brief Title: Impact of Exercise on Prognostic Biomarkers Related to Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20160604HU
Record Dates: First submitted 2018-01-04; First posted 2018-01-11 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Prostatic Neoplasm
Keywords: Prostate Cancer; Biomarkers; Exercise
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study is designed randomized controlled, 2 arm parallel group pilot study.
Masking Description: No masking was used in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-Based Exercise Program (Experimental): Participants will complete a prescribed home-based exercise program and will follow up with research staff at the UT Health San Antonio School of Nursing.
  Interventions: Other: Home-Based Exercise Program
- Waitlist-Control Group (No Intervention): Participants assigned to this group will be asked to maintain normal activity and visit the UT Health San Antonio School of Nursing for research appointments.

INTERVENTIONS:
Other: Home-Based Exercise Program — The intervention will include a combination of both aerobic and body-weight based exercises. The aerobic portion of the intervention will include 5 days of light to moderate intensity walking for 30 mins. Intensity will be set at 40-60% of the individual's heart rate reserve. The body-weight based exercises will be done 3 times a week and will consist of 3 sets of 15 reps of bodyweight squats, incline push-ups, and hip thrusts. If these exercises cannot be performed, lower intensity exercises such as sit-to-stand, wall push up and pelvic tilt can be replaced. Individuals in this group will be given a pocket guide with instructions on how to safely perform the exercises and document their completion.
  Other Names: Exercise Group
  Arms: Home-Based Exercise Program

SUMMARY:
The goal of this study is to demonstrate the impact of a home based exercise program versus wait-list control to modulate circulating prognostic biomarkers in men with prostate cancer under active surveillance.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the most common non-skin cancer effecting American males. Several reports suggest that physical activity after cancer diagnosis is associated with better cancer- specific and overall survival in individuals diagnosed with PCa. There is a growing body of evidence for lifestyle interventions that aim to promote physical activity as having the potential to counter some of the adverse effects of cancer treatments, disease progression and other health outcomes. Exercise performed 2-3 times a week has been shown to improve physical fitness, functional performance, and quality of life in men with PCa; however, few men with PCa exercise regularly and do not meet national physical activity guidelines. A potential explanation on the lack of exercise in men with PCa is the absence of a structured, home-based, exercise program. While studies have shown positive effects of exercise in men with PCa, little is known about how physical activity effects tumor physiology in men with PCa. The primary objective of this pilot study is to gather preliminary data regarding the impact of a novel, home-based exercise program on PCa biomarkers associated with recurrence and metastasis of PCa in men under active surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 40 or older
* Ambulating male
* Diagnosed with low grade prostate cancer
* Subjects willing and able to provide consent to participating in the study Exclusion Criteria
* prostatectomy
* severe cardiac disease (New York Heart Association class III or greater)
* angina
* severe osteoporosis
* uncontrolled hypertension (blood pressure > 160/95mm Hg)
* uncontrolled sinus tachycardia (> 120 beats per minute)
* uncontrolled congestive heart failure third-degree atrio-ventricular heart block, active pericarditis or myocarditis, recent embolism, thrombophlebitis, deep vein thrombosis, resting ST displacement (> 3mm), uncontrolled diabetes, uncontrolled pain, cognitive impairment, history of falls due to balance impairment or lost of consciousness,
* severe neuromusculoskeletal conditions that limit their ability to perform walking exercise (including ataxia, peripheral or sensory neuropathy, unstable bone lesion, severe arthritis, lower limb fractures within 6 months, lower limb amputation).

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants are required to have prostate cancer under active surveillance.
Enrollment: 27 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-11-19 (Actual)

PRIMARY OUTCOMES:
Change in concentration of circulating Prognostic Biomarkers | Baseline Visit, Week 12 visit, Week 18 visit and Week 24 visit.
  Analyze concentrations of Prostate-specific antigen (PSA), Prostate-specific membrane antigen (PSMA), Early prostate cancer antigen (EPCA), Urokinase plasminogen activator (uPA), and Urokinase plasminogen activator receptor (uPAR) in serum collected at each visit with research staff.

SECONDARY OUTCOMES:
Fatigue Biomarker Index | Baseline Visit, Week 12 visit, Week 18 visit and Week 24 visit.
  Analyze a novel salivary biomarker for fatigue: Measurement of the salivary biomarker, the Fatigue Biomarker Index, will be measuring the concentration of each of two peptides, GGHPPPP (SEQ ID NO:1) and ESPSLIA (SEQ ID NO:2), in a saliva sample taken from the subject then calculating the ratio of the concentration of GGHPPPP (SEQ ID NO:1) to the concentration of ESPSLIA (SEQ ID NO:2) measured according to the equation: Fatigue biomarker index (FBI)=[GGHPPPP]/[ESPSLIA]

OTHER OUTCOMES:
Improvement in Physical Function | Baseline and Week 24 visits.
  A 6-minute walk will be will be completed by participants during their initial and last appointments with research staff.
Improvement in Body Composition | Baseline visit, Week 12 visit, Week 18 visit, and Week 24 visit.
  Changes in participant's body composition will be measured at each visit with research staff.

CONTACTS AND LOCATIONS:
Overall Officials: Darpan Patel, PhD, Principal Investigator — UT Health San Antonio School of Nursing
Locations (2):
- United States (2):
  - South Texas Veterans Health Care, San Antonio, Texas
  - UT Health San Antonio School of Nursing, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galvao DA, Taaffe DR, Spry N, Joseph D, Newton RU. Combined resistance and aerobic exercise program reverses muscle loss in men undergoing androgen suppression therapy for prostate cancer without bone metastases: a randomized controlled trial. J Clin Oncol. 2010 Jan 10;28(2):340-7. doi: 10.1200/JCO.2009.23.2488. Epub 2009 Nov 30. PMID 19949016
- [Background] Keogh JW, MacLeod RD. Body composition, physical fitness, functional performance, quality of life, and fatigue benefits of exercise for prostate cancer patients: a systematic review. J Pain Symptom Manage. 2012 Jan;43(1):96-110. doi: 10.1016/j.jpainsymman.2011.03.006. Epub 2011 Jun 2. PMID 21640547
- [Background] Chan JM, Gann PH, Giovannucci EL. Role of diet in prostate cancer development and progression. J Clin Oncol. 2005 Nov 10;23(32):8152-60. doi: 10.1200/JCO.2005.03.1492. PMID 16278466
- [Background] Sonn GA, Aronson W, Litwin MS. Impact of diet on prostate cancer: a review. Prostate Cancer Prostatic Dis. 2005;8(4):304-10. doi: 10.1038/sj.pcan.4500825. PMID 16130015
- [Background] Pekmezi DW, Demark-Wahnefried W. Updated evidence in support of diet and exercise interventions in cancer survivors. Acta Oncol. 2011 Feb;50(2):167-78. doi: 10.3109/0284186X.2010.529822. Epub 2010 Nov 24. PMID 21091401
- [Background] Galvao DA, Nosaka K, Taaffe DR, Spry N, Kristjanson LJ, McGuigan MR, Suzuki K, Yamaya K, Newton RU. Resistance training and reduction of treatment side effects in prostate cancer patients. Med Sci Sports Exerc. 2006 Dec;38(12):2045-52. doi: 10.1249/01.mss.0000233803.48691.8b. PMID 17146309
- [Background] Galvao DA, Spry N, Denham J, Taaffe DR, Cormie P, Joseph D, Lamb DS, Chambers SK, Newton RU. A multicentre year-long randomised controlled trial of exercise training targeting physical functioning in men with prostate cancer previously treated with androgen suppression and radiation from TROG 03.04 RADAR. Eur Urol. 2014 May;65(5):856-64. doi: 10.1016/j.eururo.2013.09.041. Epub 2013 Oct 3. PMID 24113319
- [Background] Galvao DA, Spry N, Taaffe DR, Denham J, Joseph D, Lamb DS, Levin G, Duchesne G, Newton RU. A randomized controlled trial of an exercise intervention targeting cardiovascular and metabolic risk factors for prostate cancer patients from the RADAR trial. BMC Cancer. 2009 Dec 2;9:419. doi: 10.1186/1471-2407-9-419. PMID 19951446
- [Background] Keogh JW, Shepherd D, Krageloh CU, Ryan C, Masters J, Shepherd G, MacLeod R. Predictors of physical activity and quality of life in New Zealand prostate cancer survivors undergoing androgen-deprivation therapy. N Z Med J. 2010 Nov 5;123(1325):20-9. PMID 21317957
- [Background] Mitchell SA, Beck SL, Hood LE, Moore K, Tanner ER. Putting evidence into practice: evidence-based interventions for fatigue during and following cancer and its treatment. Clin J Oncol Nurs. 2007 Feb;11(1):99-113. doi: 10.1188/07.CJON.99-113. PMID 17441401
- [Background] Monga U, Garber SL, Thornby J, Vallbona C, Kerrigan AJ, Monga TN, Zimmermann KP. Exercise prevents fatigue and improves quality of life in prostate cancer patients undergoing radiotherapy. Arch Phys Med Rehabil. 2007 Nov;88(11):1416-22. doi: 10.1016/j.apmr.2007.08.110. PMID 17964881
- [Background] Bellizzi KM, Rowland JH, Jeffery DD, McNeel T. Health behaviors of cancer survivors: examining opportunities for cancer control intervention. J Clin Oncol. 2005 Dec 1;23(34):8884-93. doi: 10.1200/JCO.2005.02.2343. PMID 16314649
- [Background] Coups EJ, Ostroff JS. A population-based estimate of the prevalence of behavioral risk factors among adult cancer survivors and noncancer controls. Prev Med. 2005 Jun;40(6):702-11. doi: 10.1016/j.ypmed.2004.09.011. PMID 15850868
- [Background] Hansen PA, Dechet CB, Porucznik CA, LaStayo PC. Comparing eccentric resistance exercise in prostate cancer survivors on and off hormone therapy: a pilot study. PM R. 2009 Nov;1(11):1019-24. doi: 10.1016/j.pmrj.2009.09.016. PMID 19942188
- [Background] Segal RJ, Reid RD, Courneya KS, Malone SC, Parliament MB, Scott CG, Venner PM, Quinney HA, Jones LW, D'Angelo ME, Wells GA. Resistance exercise in men receiving androgen deprivation therapy for prostate cancer. J Clin Oncol. 2003 May 1;21(9):1653-9. doi: 10.1200/JCO.2003.09.534. PMID 12721238
- [Background] Obort AS, Ajadi MB, Akinloye O. Prostate-specific antigen: any successor in sight? Rev Urol. 2013;15(3):97-107. PMID 24223021
- [Background] Murphy GP, Kenny GM, Ragde H, Wolfert RL, Boynton AL, Holmes EH, Misrock SL, Bartsch G, Klocker H, Pointner J, Reissigl A, McLeod DG, Douglas T, Morgan T, Gilbaugh J Jr. Measurement of serum prostate-specific membrane antigen, a new prognostic marker for prostate cancer. Urology. 1998 May;51(5A Suppl):89-97. doi: 10.1016/s0090-4295(98)00082-x. PMID 9610563
- [Background] Zhao Z, Ma W, Zeng G, Qi D, Ou L, Liang Y. Preoperative serum levels of early prostate cancer antigen (EPCA) predict prostate cancer progression in patients undergoing radical prostatectomy. Prostate. 2012 Feb;72(3):270-9. doi: 10.1002/pros.21428. Epub 2011 May 31. PMID 21630293
- [Background] Gupta A, Lotan Y, Ashfaq R, Roehrborn CG, Raj GV, Aragaki CC, Montorsi F, Shariat SF. Predictive value of the differential expression of the urokinase plasminogen activation axis in radical prostatectomy patients. Eur Urol. 2009 May;55(5):1124-33. doi: 10.1016/j.eururo.2008.06.054. Epub 2008 Jun 23. PMID 18585843
- [Background] Shariat SF, Roehrborn CG, McConnell JD, Park S, Alam N, Wheeler TM, Slawin KM. Association of the circulating levels of the urokinase system of plasminogen activation with the presence of prostate cancer and invasion, progression, and metastasis. J Clin Oncol. 2007 Feb 1;25(4):349-55. doi: 10.1200/JCO.2006.05.6853. PMID 17264329
- [Background] Shariat SF, Semjonow A, Lilja H, Savage C, Vickers AJ, Bjartell A. Tumor markers in prostate cancer I: blood-based markers. Acta Oncol. 2011 Jun;50 Suppl 1(Suppl 1):61-75. doi: 10.3109/0284186X.2010.542174. PMID 21604943
- [Background] Chen CL, Mahalingam D, Osmulski P, Jadhav RR, Wang CM, Leach RJ, Chang TC, Weitman SD, Kumar AP, Sun L, Gaczynska ME, Thompson IM, Huang TH. Single-cell analysis of circulating tumor cells identifies cumulative expression patterns of EMT-related genes in metastatic prostate cancer. Prostate. 2013 Jun;73(8):813-26. doi: 10.1002/pros.22625. Epub 2012 Dec 31. PMID 23280481
- [Background] Gupta D, Lis CG, Grutsch JF. The relationship between cancer-related fatigue and patient satisfaction with quality of life in cancer. J Pain Symptom Manage. 2007 Jul;34(1):40-7. doi: 10.1016/j.jpainsymman.2006.10.012. Epub 2007 May 25. PMID 17532179
- [Background] Campos MPO, Hassan BJ, Riechelmann R, Del Giglio A. Cancer-related fatigue: a practical review. Ann Oncol. 2011 Jun;22(6):1273-1279. doi: 10.1093/annonc/mdq458. Epub 2011 Feb 16. PMID 21325448
- [Background] Michael DJ, Daugherty S, Santos A, Ruby BC, Kalns JE. Fatigue biomarker index: an objective salivary measure of fatigue level. Accid Anal Prev. 2012 Mar;45 Suppl:68-73. doi: 10.1016/j.aap.2011.09.029. Epub 2011 Oct 10. PMID 22239935
- [Background] Kalns J, Baskin J, Reinert A, Michael D, Santos A, Daugherty S, Wright JK. Predicting success in the tactical air combat party training pipeline. Mil Med. 2011 Apr;176(4):431-7. doi: 10.7205/milmed-d-10-00110. PMID 21539166
- [Background] Zoukhri D, Kublin CL. Impaired neurotransmitter release from lacrimal and salivary gland nerves of a murine model of Sjogren's syndrome. Invest Ophthalmol Vis Sci. 2001 Apr;42(5):925-32. PMID 11274068
- [Background] Lubeck DP, Litwin MS, Henning JM, Stoddard ML, Flanders SC, Carroll PR. Changes in health-related quality of life in the first year after treatment for prostate cancer: results from CaPSURE. Urology. 1999 Jan;53(1):180-6. doi: 10.1016/s0090-4295(98)00408-7. PMID 9886609

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT03397030/Prot_SAP_000.pdf